CLINICAL TRIAL: NCT07211360
Title: Integrated PET/MR Imaging With Amino Acid Radiotracers in the Evaluation of Brain Neoplasms: Assessing Diagnostic Accuracy and Therapeutic Response
Acronym: PETMR_ATHENA02
Status: Not yet recruiting | Type: Observational
Sponsor: IRCCS San Raffaele (Other)
Responsible Party: Principal Investigator, Chiti Arturo, Prof., IRCCS San Raffaele
Other Study IDs: 3426
Record Dates: First submitted 2025-08-06; First posted 2025-10-07 (Actual); Last update posted 2025-10-07 (Actual); Status verified 2025-09

CONDITIONS: Primary and Secondary Brain Tumors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cohort A: Adult patients with primary or secondary brain tumors undergoing neuro-oncological therapy, presenting with lesions suspected to be either disease progression or post-treatment changes
- cohort B: Adult patients with a first diagnosis of primary or secondary brain tumor.

SUMMARY:
Evaluation of the diagnostic and prognostic role of PET with Amino Acid Radiotracers associated with simultaneous acquisition of MRI with administration of paramagnetic contrast medium based on Gadobutrol in assessing diagnostic accuracy and therapeutic response in adult individuals affected by primary and secondary brain tumors. This is a purely observational study that does not introduce any procedures beyond those already scheduled as part of routine clinical practice. All imaging procedures and clinical assessments will be performed exclusively within the standard care pathway. This study will analyze two cohorts of patients:

1. Cohort A: Adult patients with primary or secondary brain tumors undergoing neuro-oncological therapy, presenting with lesions suspected to be either disease progression or post-treatment changes.

2. Cohort B: Adult patients with a first diagnosis of primary or secondary brain tumor.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-99.
2. Diagnosis of primary or secondary brain tumors.
3. Development of suspected lesions on MRI following treatment, with dimensions greater than one centimeter.
4. Ability to undergo PET/MRI imaging sessions.
5. Availability of clinical and follow-up data for correlation with imaging findings
6. Signed informed consent from the patient

Exclusion Criteria:

.Patients under 18 years of age. 2.Absence of a confirmed diagnosis of primary or secondary brain tumors. 3.Lesions on MRI with dimensions smaller than one centimeter. 4.Inability to undergo PET/MRI imaging sessions (e.g., due to medical conditions such as pregnancy, allergies to contrast agents, or presence of incompatible implants or devices) 5.Unavailability of clinical and follow-up data for correlation with imaging findings.

6.Patients who are unable or unwilling to provide signed informed consent.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult individuals affected by primary and secondary brain tumors.
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-10-01 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2031-09 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of PET/MRI | Conducted at approximately the end of the planned treatment course.
  Diagnostic accuracy of PET/MRI measured with sensitivity, specificity (calculated from the contingency table as follows: Sensitivity = True Positives / (True Positives + False Negatives) and Specificity True Negatives / (True Negatives + False Positives), positive and negative predicted value using clinical radiological or histopathology outcomes collected during standard clinical practice.
Clinical-radiological outcome | Conducted at approximately the end of the planned treatment course
  it will be defined as disease progression if serial imaging shows a >25% increase in lesion size or the appearance of new lesions, according to RANO or BTRADS criteria.
Histopathology outcome | Conducted at approximately the end of the planned treatment course
  it involves tissue biopsy results confirmed by pathology reports